CLINICAL TRIAL: NCT02182193
Title: Safety and Relative Bioavailability of a Single Dose of 150 mg BIBF 1120 Administered as Soft Gelatine Capsules Charge 1 Compared to BIBF 1120 Soft Gelatine Capsules Charge 2 Compared to BIBF 1120 Administered as Drinking Solution Following Oral Administration to Healthy Male Volunteers in an Open, Randomised, Intra-individual, Crossover Comparison Design
Brief Title: Safety and Relative Bioavailability of BIBF 1120 Soft Gelatine Capsules Charge 1, BIBF 1120 Soft Gelatine Capsules Charge 2 and BIBF 1120 Drinking Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1199.21
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- BIBF 1120 capsules charge 1 (Experimental)
  Interventions: Drug: BIBF 1120 capsules charge 1
- BIBF 1120 capsules charge 2 (Experimental)
  Interventions: Drug: BIBF 1120 capsules charge 2
- BIBF 1120 drinking solution (Active Comparator)
  Interventions: Drug: BIBF 1120 drinking solution

INTERVENTIONS:
Drug: BIBF 1120 capsules charge 1
  Arms: BIBF 1120 capsules charge 1
Drug: BIBF 1120 capsules charge 2
  Arms: BIBF 1120 capsules charge 2
Drug: BIBF 1120 drinking solution
  Arms: BIBF 1120 drinking solution

SUMMARY:
To assess pharmacokinetics and the relative bioavailability of a single dose of BIBF 1120 soft gelatine capsule charge 1 vs. BIBF 1120 soft gelatine capsule charge 2 vs BIBF 1120 drinking solution in healthy male subjects respectively. To establish an in-vitro-in-vivo correlation (IVIVC) for oral soft gelatine capsules with 150 mg BIBF 1120 in healthy male volunteers (if feasible)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects as determined by results of screening
2. Signed written informed consent in accordance with GCP and local legislation
3. Age ≥21 and ≤55 years
4. Body Mass Index ≥18.5 kg/m2 and ≤29.9 kg/m2

Exclusion Criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
2. History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
3. History of relevant orthostatic hypotension, fainting spells and blackouts
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy or its excipients) which is deemed relevant to the trial as judged by the investigator
7. History of any bleeding disorder including prolonged or habitual bleeding, other hematologic disease or cerebral bleeding (e.g. after a car accident) or commotio cerebri
8. Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
9. Use of any drugs which might influence the results of the trial within 14 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within 2 months prior to administration or during trial
11. Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
12. Alcohol abuse (> 60 g/day)
13. Drug abuse
14. Blood donation (more than 150 mL within 4 weeks prior to administration or during the trial)
15. Excessive physical activities within 5 days prior to administration or during the trial
16. Any laboratory value outside the reference range that is of clinical relevance
17. Female gender
18. Male subjects refuse to minimize the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than 3 months prior to dosing, barrier contraception or a medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intra-uterine device, tubal ligation, hormonal contraceptive since at least two months and diaphragm with spermicide

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2006-09; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve of the analyte from zero time (pre-dose) extrapolated to infinity (AUC0-∞) | 1 h pre dose and up to 48 h after drug administration
Individual maximum observed concentrations of the analyte in plasma (Cmax) | 1 h pre dose and up to 48 h after drug administration

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve of the analyte over the time interval from time zero (pre-dose) to 24 hours (AUC0-24) | 1 h pre dose and up to 24 h after drug administration
time from dosing to the maximum concentration of the analyte in plasma (tmax) | 1 h pre dose and up to 48 h after drug administration
Terminal rate constant in plasma (λz) | 1 h pre dose and up to 48 h after drug administration
Terminal half-life of the analyte in plasma (t1/2) | 1 h pre dose and up to 48 h after drug administration
Mean residence time of the analyte in the body after oral administration (MRTpo) | 1 h pre dose and up to 48 h after drug administration
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F) | 1 h pre dose and up to 48 h after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | 1 h pre dose and up to 48 h after drug administration
Change in vital signs (blood pressure, pulse rate) | Baseline, up to 24 hours after drug administration
Change in routine laboratory values | pre-dose, up to 48 hours after drug administration
Change in ECG | pre-dose, 4 hours after drug administration, day 32
Occurrence of adverse events | up to 32 days after drug administration
Assessment of tolerability by investigator on a 4 point scale | 48 hours after drug administration